CLINICAL TRIAL: NCT01619423
Title: A Double Blinded Randomised Three Armed Phase II Trial of PledOx in Two Different Doses in Combination With FOLFOX6 Compared to Placebo + FOLFOX6 in Patients With Advanced Metastatic Colorectal (Stage IV) Cancer
Brief Title: A Trial of PledOx + FOLFOX6 Compared to Placebo + FOLFOX6 in Patients With Metastatic Colorectal Cancer
Acronym: PLIANT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Egetis Therapeutics (Industry)
Collaborators: Pharma Consulting Group AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PP095, (PLIANT); 2012-001367-76 (EudraCT Number)
Record Dates: First submitted 2012-05-25; First posted 2012-06-14 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Advanced Metastatic (Stage IV) Colorectal Cancer
Keywords: Metastatic colorectal cancer; stage IV; FOLFOX6; Chemotherapy; PledOx; Mangafodipir; Febrile neutropenia; Oxidative stress; Antioxidant; neutropenia; neuropathy
MeSH Terms: conditions — Colorectal Neoplasms; Febrile Neutropenia; Neutropenia | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is a three arm study, however, we changed the high dose in the secord part of the study, from 10 micromol/kg (part 2a) to 5 mictomol/kg (part 2b)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FOLFOX6 + PledOx 2 µmol/kg (Active Comparator): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  Interventions: Drug: PledOx (2 µmol/kg)
- FOLFOX6 + PledOx 5 µmol/kg (Active Comparator): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  Interventions: Drug: PledOx (5 µmol/kg)
- FOLFOX6 + PledOx 10 µmol/kg (Active Comparator): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  Interventions: Drug: PledOx (10 µmol/kg)
- FOLFOX6 + 0,9% NaCl (Placebo Comparator): Placebo= 0.9% NaCl; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  Interventions: Drug: Placebo (0,9% NaCl)

INTERVENTIONS:
Drug: PledOx (2 µmol/kg) — PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
  Other Names: Calmangafodipir
  Arms: FOLFOX6 + PledOx 2 µmol/kg
Drug: PledOx (5 µmol/kg) — PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles
  Other Names: Calmangafodipir
  Arms: FOLFOX6 + PledOx 5 µmol/kg
Drug: PledOx (10 µmol/kg) — PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles
  Other Names: Calmangafodipir
  Arms: FOLFOX6 + PledOx 10 µmol/kg
Drug: Placebo (0,9% NaCl) — Placebo (0,9% NaCl) is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
  Other Names: Sodium chloride
  Arms: FOLFOX6 + 0,9% NaCl

SUMMARY:
The present trial is designed to determine whether pre-treatment with PledOx lowers the frequency and severity of side effects from FOLFOX6 administration in patients with metastatic colorectal cancer.

The efficacy of PledOx will be assessed when added to FOLFOX6 chemotherapy as first line treatment of metastatic colorectal cancer.

This study was performed in multiple parts/phases. Part 1 was an open dose-escalation study with the doses 2, 5 and 10 micromol/kg of calmangafodipir. No study outcomes were planned for this part. In part 2a, participants randomly received either Placebo, 2 or 10 micromol/kg of calmangafodipir. In part 2b, participants randomly received either Placebo, 2 or 5 micromol/kg of calmangafodipir. The overall intent of the study was to compare the effect of antioxidant agent PledOx against placebo in one of three different doses/combinations (2 micromol/kg, 5/10 micromol/kg, 2/5/10 micromol/kg vs. placebo, in the first 8 cycles of FOLFOX6 treatment

DETAILED DESCRIPTION:
Globally, nearly 800 000 colorectal cancers are believed to occur annually. Approximately about half of the patients with colorectal cancer develop metastatic disease. These patients are often offered chemotherapy with the FOLFOX6 regimen (FOL = FOLic acid; F = Fluorouracil (5-FU); OX = OXaliplatin) The use of FOLFOX6 is, however, hampered by a high incidence and severity of adverse reactions.

In the current trial patients will receive the antioxidant agent PledOx in one of two different doses, or placebo, in the first 8 cycles of FOLFOX6 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced metastatic colorectal (stage IV) cancer verified by biopsy
* Patients may have received up to three previous treatment lines of chemotherapy, which may include fluoropyrimidine, irinotecan and targeted therapies. The last dose of antitumor drug must be given at least 4 weeks prior to inclusion and all toxicity (except alopecia and fatigue) resolved. Patients may also be chemotherapy-naïve, have received prior adjuvant treatment but no previous treatment with oxaliplatin
* CT-scan or MRI of thorax, abdomen and pelvis; within ≤4 weeks before start of chemotherapy
* Evaluable disease and one measurable site of disease according to RECIST 1.1 criteria (at least 10mm for CT-scan or MRI)
* Neurological examination with no significant pathological findings
* ≥18 years
* WHO performance status 0≤2 and Life expectancy ≥ 3 months
* Adequate haematological function, Hb ≥ 100 g/L, ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L
* Adequate renal and hepatic functions: creatinine clearance >50 cc/min, total bilirubin ≤ 1.5 times ULN, ASAT and ALAT ≤ 3 times ULN (ASAT and ALAT ≤ 5 times ULN in case of liver metastases)
* INR ≤1.5 times ULN, unless receiving therapeutic anticoagulation
* Negative pregnancy test for females of child-producing potential
* Written informed consent given

Exclusion Criteria:

* Tumours other than colorectal adenocarcinomas (within the previous 5 years) except for curatively treated non melanoma skin cancer or in situ carcinoma of the cervix
* Evidence of central nervous system metastases
* Unresolved bowel obstruction or sub-obstruction, uncontrolled Crohn's disease or ulcerative colitis
* History of cardiac disease with a New York Heart Association (NYHA) Class II or greater congestive heart failure, myocardial infarction or unstable angina in the past six (6) months prior to Day 1 of treatment and serious arrhythmias requiring medication for treatment
* Prolonged QTC interval >450 msec
* Known history of stroke or cerebrovascular accident in the past six (6) months
* Severe diarrhoea
* Chronic infection or uncontrolled serious illness causing immunodeficiency
* Any uncontrolled serious illness or medical condition
* Received mangafodipir at any time
* Welders, mine workers or other workers in occupations (current or past) where high manganese exposure is likely
* Pre-existing neurodegenerative disease (Parkinson's, Alzheimer's, Huntington's etc.) or neuromuscular disorder (Multiple sclerosis, Amyotrophic lateral sclerosis, Polio, hereditary neuromuscular disease)
* Major psychiatric disorder (major depression, psychosis)
* Participation in another clinical study with an investigational medicinal product within 1 month prior to inclusion.
* Blood manganese concentration values >18.3 μg/L at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bengtson, Study Director — Egetis Therapeutics
Locations (33):
- United States (6):
  - Moores UCSD Cancer Center, La Jolla, California
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Associates in Oncology & Hematology, Chattanooga, Tennessee
  - Wellmont Medical Associates Oncology and Hematology, Kingsport, Tennessee
  - The University of Texas, Health Science Center at San Antonio, San Antonio, Texas
  - Benaroya Research Institute @ Virginia Mason, Seattle, Washington
- Bulgaria (5):
  - Complex Oncology Center-Plovdiv EOOD, Department of Medical Oncology and oncology diseases in gastroenterology, Plovdiv
  - Complex Oncology Center-Shumen EOOD, Department of Medical Oncology, Shumen
  - MHAT "Serdika" EOOD, Department of Medical Oncology, Sofia
  - UMHAT "Tzaritza Joanna-ISUL" EAD, Clinic of Medical Oncology, Sofia
  - SHATO EAD, Sofia, Clinic of Chemotherapy, Sofia
- Denmark (2):
  - Aalborg University Hospital, Dept of Oncology, Clinical Research Unit, Aalborg
  - Odense Universitetshospital, Klinisk Forsknings Enhed, Onkologisk Afdelig R, Odense
- Georgia (5):
  - LTD Clinic Medina, Batumi
  - Resaerch Institte of Clinical Medicine, Tbilisi
  - JSC "Neo Medi", Tbilisi
  - LTD " High Technology Medical Center University Clinic", Tbilisi
  - S. Khechinashvili University Hospital, Tbilisi
- Germany (3):
  - St. Josef-Hospital -Universitätsklinik Ruhr-Universität Bochum, Leitende Ärztin der Abt. für Hämatologie und Onkologie, Medizinische Klinik I, Bochum
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie -Onkologie, Dresden
  - HELIOS Klinikum Wuppertal, Klinik für Hämatologie und Onkologie, Wuppertal
- Portugal (3):
  - Centro Hospitalar do Baixo Vouga, E.P.E. (Hospital Infante D. Pedro), Oncologia Médica, Aveiro
  - Hospital de Braga, Oncologia Médica, Braga
  - Instituto Português de Oncologia do Porto, Francisco Gentil, E.P.E., Oncologia Médica, Porto
- Serbia (4):
  - Institute for Oncology and Radiology of Serbia, Clinic for Medical Oncology, Belgrade
  - Military Medical Academy, Gastroenterology department, Belgrade
  - Clinical Hospital Center Zemun, Insitute for Oncology, Belgrade
  - Clinical Center Kragujevac, Center for Oncology, Kragujevac
- Sweden (5):
  - Gävle sjukhus, Oncology unit, Gävle
  - Sahlgrenska/Östra sjukhuset, Gothenburg
  - Universitetssjukhuset i Linköping, Linköping
  - Karolinska Sjukhuset, Stockholm
  - Akademiska Sjukhuset, Uppsala

REFERENCES:
- [Result] Glimelius B, Manojlovic N, Pfeiffer P, Mosidze B, Kurteva G, Karlberg M, Mahalingam D, Buhl Jensen P, Kowalski J, Bengtson M, Nittve M, Nasstrom J. Persistent prevention of oxaliplatin-induced peripheral neuropathy using calmangafodipir (PledOx(R)): a placebo-controlled randomised phase II study (PLIANT). Acta Oncol. 2018 Mar;57(3):393-402. doi: 10.1080/0284186X.2017.1398836. Epub 2017 Nov 15. PMID 29140155

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 186 participants were enrolled and 186 started the study, however, two patients had too high basal manganese levels (detected after first treatment cycle) and were excluded from further treatment (screening failures) but are part of the safety population. 184 patients are part of the treatment population (11 in part 1 and 173 in part 2)
Groups:
- FOLFOX6 + 0,9% NaCl (Part 2a+2b): Placebo= 0.9% NaCl; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  Placebo (0,9% NaCl): Placebo (0,9% NaCl) is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
- FOLFOX6 + PledOx 2 µmol/kg (Part 1, 2a+2b): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  PledOx (2 µmol/kg): PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
- FOLFOX6 + PledOx 5 µmol/kg (Part 1, 2b): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  PledOx (5 µmol/kg): PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
- FOLFOX6 + PledOx 10 µmol/kg (Part 1, 2a): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  PledOx (10 µmol/kg): PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
Period: Part 1 (Dose Escalation)
Arm/Group | FOLFOX6 + 0,9% NaCl (Part 2a+2b) | FOLFOX6 + PledOx 2 µmol/kg (Part 1, 2a+2b) | FOLFOX6 + PledOx 5 µmol/kg (Part 1, 2b) | FOLFOX6 + PledOx 10 µmol/kg (Part 1, 2a)
Started | 0 | 5 | 3 | 5
Completed | 0 | 3 | 3 | 5
Not Completed | 0 | 2 | 0 | 0
Not completed — High basal Mn | 0 | 2 | 0 | 0
Period: Part 2a
Arm/Group | FOLFOX6 + 0,9% NaCl (Part 2a+2b) | FOLFOX6 + PledOx 2 µmol/kg (Part 1, 2a+2b) | FOLFOX6 + PledOx 5 µmol/kg (Part 1, 2b) | FOLFOX6 + PledOx 10 µmol/kg (Part 1, 2a)
Started | 15 | 13 | 0 | 11
Completed | 15 | 13 | 0 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Part 2b
Arm/Group | FOLFOX6 + 0,9% NaCl (Part 2a+2b) | FOLFOX6 + PledOx 2 µmol/kg (Part 1, 2a+2b) | FOLFOX6 + PledOx 5 µmol/kg (Part 1, 2b) | FOLFOX6 + PledOx 10 µmol/kg (Part 1, 2a)
Started | 45 | 44 | 45 | 0
Completed | 45 | 44 | 45 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Although no pre-specified Outcome Measures were performed on participants in Part 1, however, baseline data for all 186 participants is reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFOX6 + 0,9% NaCl (Part 2a+2b) | FOLFOX6 + PledOx 2 µmol/kg (Part 1, 2a+2b) | FOLFOX6 + PledOx 5 µmol/kg (Part 1, 2b) | FOLFOX6 + PledOx 10 µmol/kg (Part 1, 2a) | Total
Number analyzed (Participants) | 60 | 62 | 48 | 16 | 186
Age, Continuous [Mean (Full Range); unit: years] | 62 [41 to 80] | 63.5 [42 to 83] | 62.6 [38 to 82] | 61.3 [35 to 80] | 62.6 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 26 | 7 | 125
  Male | 14 | 16 | 22 | 9 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 58 | 61 | 45 | 16 | 180
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Neuropathy Grade 2 or Higher (According to the Oxaliplatin Specific Sanofi Scale (OSSS) Criteria Related Paraesthesia/Dysaesthesia)
Description: Percentage of patients, over cycle 1 to 8, with neuropathy grade 2 or higher (according to the Oxaliplatin Specific Sanofi Scale (OSSS) criteria related paraesthesiae/dysaesthesiae)
Time Frame: Every second week during cycle 1-8, for up to 16 weeks
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Control group
- FOLFOX6 + PledOx 5+10 µmol/kg: PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  Combined PledOx (5 and 10 µmol/kg groups): PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
- FOLFOX6 + PledOx 2+5+10 µmol/kg: PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  Combined PledOx (2, 5 and 10 µmol/kg groups): PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
Arm/Group | Placebo | FOLFOX6 + PledOx 2 µmol/kg | FOLFOX6 + PledOx 5+10 µmol/kg | FOLFOX6 + PledOx 2+5+10 µmol/kg
Number analyzed (Participants) | 60 | 57 | 56 | 113
Participants | 14 | 11 | 6 | 17
Statistical Analysis 1: Comparison: Placebo vs FOLFOX6 + PledOx 2 µmol/kg; Test type: Superiority; p = 0.31, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.78, 10% CI 1-sided [upper limit 1.5]
Statistical Analysis 2: Comparison: Placebo vs FOLFOX6 + PledOx 5+10 µmol/kg; Test type: Superiority; p = 0.15, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.55, 10% CI 1-sided [upper limit 1.16]
Statistical Analysis 3: Comparison: Placebo vs FOLFOX6 + PledOx 2+5+10 µmol/kg; Test type: Superiority; p = 0.16, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.62, 10% CI 1-sided [upper limit 1.14]

ADVERSE EVENTS:
Time Frame: 30 days after last treatment for newly occuring AE:s and until resolution for ongoing, up to 2 years from baseline
Groups:
- Part 1 (Dose Escalation): Part 1 is an open dose-escalation part with the doses 2, 5 and 10 µmol/kg of PledOx with the active ingridient calmangafodipir
- FOLFOX6 + PledOx 2 µmol/kg (Part 2a+2b): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  PledOx (2 µmol/kg): PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
- FOLFOX6 + PledOx 5 µmol/kg (Part 2b): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  PledOx (5 µmol/kg): PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
- FOLFOX6 + PledOx 10 µmol/kg (Part 2a): PledOx active ingredient= Calmangafodipir; FOLFOX6=Combination of FOLinic Acid, 5-Fluorouracil (5-FU), and Oxaliplatin.
  PledOx (10 µmol/kg): PledOx is administered intravenously for up to 5 minutes, about 10 min prior to start of FOLFOX6 chemotherapy which will be administered day 1 and 2 every second week for up to 8 cycles.
Arm/Group | FOLFOX6 + 0,9% NaCl (Part 2a+2b) | Part 1 (Dose Escalation) | FOLFOX6 + PledOx 2 µmol/kg (Part 2a+2b) | FOLFOX6 + PledOx 5 µmol/kg (Part 2b) | FOLFOX6 + PledOx 10 µmol/kg (Part 2a)
All-Cause Mortality (participants affected / at risk) | 2/60 | 0/13 | 1/57 | 1/45 | 1/11
Serious Adverse Events (participants affected / at risk) | 6/60 | 2/13 | 7/57 | 3/45 | 2/11
Other Adverse Events (participants affected / at risk) | 49/60 | 10/13 | 45/57 | 35/45 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX6 + 0,9% NaCl (Part 2a+2b) (N=60) | Part 1 (Dose Escalation) (N=13) | FOLFOX6 + PledOx 2 µmol/kg (Part 2a+2b) (N=57) | FOLFOX6 + PledOx 5 µmol/kg (Part 2b) (N=45) | FOLFOX6 + PledOx 10 µmol/kg (Part 2a) (N=11)
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Staphyloccocal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hypersensitivty (Immune system disorders) | 1 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestine obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0
Cheast pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Stoma site hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Central venous catherization (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Stoma closure (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX6 + 0,9% NaCl (Part 2a+2b) (N=60) | Part 1 (Dose Escalation) (N=13) | FOLFOX6 + PledOx 2 µmol/kg (Part 2a+2b) (N=57) | FOLFOX6 + PledOx 5 µmol/kg (Part 2b) (N=45) | FOLFOX6 + PledOx 10 µmol/kg (Part 2a) (N=11)
Blood and lymphatic system disorder (Blood and lymphatic system disorders) | 49 | 10 | 45 | 35 | 9
Nervous system disorder (Nervous system disorders) | 47 | 7 | 44 | 32 | 8
Gastrointestinal disorder (Gastrointestinal disorders) | 36 | 9 | 31 | 32 | 8
General disorders (General disorders) | 35 | 2 | 24 | 28 | 2
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 19 | 5 | 18 | 11 | 2
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 7 | 7 | 0
Skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 7 | 2 | 7 | 3 | 2
Infections and infestations (Infections and infestations) | 4 | 2 | 6 | 3 | 0
Investigations (Investigations) | 6 | 1 | 5 | 5 | 2
Musculosceletal and connective tissue (Musculoskeletal and connective tissue disorders) | 7 | 2 | 3 | 6 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The pre-specified statistical analysis plan (SAP) states; if the primary outcome meassure failed, then all additional outcome measures are considered exploratory. A selected number of the exploratory outcomes are presented in the linked publication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No